CLINICAL TRIAL: NCT01475981
Title: Randomized,Double-blind,Placebo-controlled,Ascending Dose Part Evaluating Safety,Tolerability and Pharmacokinetics (PK) of JTK-853 (Fasted/Fed) and Randomized,Open-label,Crossover Part Evaluating Food Effect on PK in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics Study Assessing Ascending Single Oral JTK-853 Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK853-U-09-001
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: JTK-853; single dose
MeSH Terms: interventions — JTK-853

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Dose 1 JTK-853 (fasted condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 2 JTK-853 (fasted condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 3 JTK-853 (fasted condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 2 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 3 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 4 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 5 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 6 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 7 JTK-853 (fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 5 JTK-853 (high-fat fed condition) (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: JTK-853 or Placebo

INTERVENTIONS:
Drug: JTK-853 or Placebo — Tablets, single dose, fasted, fed or high-fat fed condition

SUMMARY:
The purpose of this study was to determine the safety, tolerability and pharmacokinetics of ascending single oral doses of JTK-853 administered under fasted or fed conditions in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) of 18-30 kg/m2 (inclusive)
2. Non-smokers or subjects who have stopped smoking at least 6 months prior to the Screening Visit

Exclusion Criteria:

1. History or presence of cardiac disease, including a family history of long-QT syndrome or unexplained sudden death
2. Have used any prescription medication, herbal product, or over-the-counter (OTC) medication (except acetaminophen), within 4 weeks prior to the Day before dosing

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 1 week
Maximum concentration (Cmax) of JTK-853 and metabolite M2 | 1 week
Time to reach peak or maximum concentration following drug administration (tmax) for JTK-853 and metabolite M2 | 1 week
Area under the concentration-time curve from the time of dosing to the last quantifiable time point (AUClast) for JTK-853 and metabolite M2 | 1 week
Area under the concentration-time curve from the time of dosing to infinity (AUCinf) for JTK-853 and metabolite M2 | 1 week
Elimination half-life associated with the terminal slope (λz) of a semilogarithmic concentration-time curve (t1/2) for JTK-853 and metabolite M2 | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Hoshino, D.V.M, Study Director — Akros Pharma Inc.
Locations (1):
- PPD, Phase I Clinic, Austin, Texas, United States